CLINICAL TRIAL: NCT02861573
Title: Phase Ib/II Trial of Pembrolizumab (MK-3475) Combination Therapies in Metastatic Castration-Resistant Prostate Cancer (mCRPC) (KEYNOTE-365)
Brief Title: Study of Pembrolizumab (MK-3475) Combination Therapies in Metastatic Castration-Resistant Prostate Cancer (MK-3475-365/KEYNOTE-365)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-365; KEYNOTE-365 (Other: MSD); MK-3475-365 (Other: MSD); 2023-506987-15-00 (Registry Identifier: EU CT); U1111-1294-7577 (Registry Identifier: UTN); 2016-002312-41 (EudraCT Number)
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer; mCRPC; PD1; PD-1; PDL1; PD-L1
MeSH Terms: interventions — pembrolizumab; olaparib; Docetaxel; Prednisone; enzalutamide; Dexamethasone; Abiraterone Acetate; lenvatinib; Carboplatin; Etoposide; belzutifan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Pembrolizumab+Olaparib (Experimental): Participants with adenocarcinoma (AC) mCRPC in Cohort A will receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week dosing cycle (Q3W) and olaparib 400 mg capsules or 300 mg tablets by mouth (PO) twice a day (BID) continuously from Day 1 of Cycle 1. Treatment with pembrolizumab will continue until progression or a maximum of 35 treatment cycles (up to 2 years). Treatment with olaparib will continue until progression. Participants who must discontinue 1 of the 2 drugs in the combination due to adverse events may continue the study with the other combination drug.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Olaparib 400 mg; Drug: Olaparib 300 mg
- Pembrolizumab+Docetaxel+Prednisone (Experimental): Participants with AC mCRPC in Cohort B will receive pembrolizumab 200 mg IV on Day 1 Q3W, docetaxel 75 mg/m^2 IV on Day 1 Q3W, and prednisone 5 mg tablet PO BID continuously from Day 1 of Cycle 1. Participants will only be permitted to receive a maximum of 10 cycles of docetaxel and prednisone. Treatment with pembrolizumab will continue for a maximum of 35 cycles (up to 2 years) or until progression. Participants who must discontinue 1 of the 2 drugs due to adverse events in the combination may continue the study with the other combination drug.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Docetaxel 75 mg/m^2; Drug: Prednisone 5 mg; Other: Dexamethasone 8 mg
- Pembrolizumab+Enzalutamide (Experimental): Participants with AC mCRPC in Cohort C will receive pembrolizumab 200 mg IV on Day 1 Q3W and enzalutamide 160 mg PO every day (QD) continuously from Day 1 of Cycle 1. Treatment with pembrolizumab will continue until progression or a maximum of 35 treatment cycles (up to 2 years). Treatment with enzalutamide will continue until progression. Participants who must discontinue 1 of the 2 drugs in the combination due to adverse events may continue the study with the other combination drug.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Enzalutamide 160 mg
- Pembrolizumab+Abiraterone+Prednisone (Experimental): Participants with AC mCRPC in Cohort D will receive pembrolizumab 200 mg IV on Day 1 Q3W, abiraterone acetate 1000 mg PO QD and prednisone 5 mg tablet PO BID continuously from Day 1 of Cycle 1. Treatment with pembrolizumab will continue for a maximum of 35 cycles (up to 2 years) or until progression. Participants who must discontinue 1 of the 2 drugs due to adverse events in the combination may continue the study with the other combination drug.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Prednisone 5 mg; Drug: Abiraterone acetate 1000 mg
- Pembrolizumab+Lenvatinib: AC (Experimental): Participants with AC mCRPC in Cohort E will receive pembrolizumab 200 mg IV on Day 1 Q3W, and lenvatinib 20 mg PO QD continuously from Day 1 of Cycle 1. Treatment with pembrolizumab will continue for a maximum of 35 cycles (up to 2 years) or until progression. Participants who must discontinue 1 of the 2 drugs due to adverse events in the combination may continue the study with the other combination drug.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Lenvatinib
- Pembrolizumab+Lenvatinib:t-NE (Experimental): Participants with neuroendocrine (t-NE) mCRPC in Cohort F will receive pembrolizumab 200 mg IV on Day 1 Q3W, and lenvatinib 20 mg PO QD continuously from Day 1 of Cycle 1. Treatment with pembrolizumab will continue for a maximum of 35 cycles (up to 2 years) or until progression. Participants who must discontinue 1 of the 2 drugs due to adverse events in the combination may continue the study with the other combination drug.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Lenvatinib
- Pembrolizumab/Vibostolimab coformulation (Experimental): Participants with AC mCRPC in Cohort G will receive a coformulation fixed dose combination of 200 mg pembrolizumab and 200 mg vibostolimab (MK-7684) Q3W IV from Day 1 of Cycle 1. Treatment will continue for a maximum of 35 cycles (up to 2 years) or until progression.
  Interventions: Biological: Pembrolizumab/Vibostolimab coformulation
- Pembrolizumab/Vibostolimab coformulation:t-NE (Experimental): Participants with t-NE mCRPC in Cohort H will receive a coformulation fixed dose combination of 200 mg pembrolizumab and 200 mg vibostolimab (MK-7684) Q3W IV from Day 1 of Cycle 1. Treatment will continue for a maximum of 35 cycles (up to 2 years) or until progression.
  Interventions: Biological: Pembrolizumab/Vibostolimab coformulation
- Pembrolizumab+Carboplatin+Etoposide (Experimental): Participants with neuroendocrine mCRPC in Cohort I Arm 1 will receive pembrolizumab 200 mg IV on Day 1 Q3W + carboplatin titrated to an area under the plasma drug concentration-time curve [AUC] 5 IV on Day 1 Q3W + etoposide 100 mg/m^2 IV on Days 1, 2, and 3 Q3W. Treatment with pembrolizumab will continue for a maximum of 35 cycles (up to 2 years) or until progression. Treatment with carboplatin+etoposide will continue for a maximum of 4 cycles (up to 2.8 months). Participants who must discontinue 1 or 2 of the 3 drugs due to adverse events in the combination may continue the study with the other combination drug/drugs.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Carboplatin; Drug: Etoposide
- Carboplatin+Etoposide (Experimental): Participants with neuroendocrine mCRPC in Cohort I Arm 2 will receive carboplatin titrated to an area under the plasma drug concentration-time curve [AUC] 5 IV on Day 1 Q3W + etoposide 100 mg/m^2 IV on Days 1, 2, and 3 Q3W. Treatment will continue for a maximum of 35 cycles (up to 2 years) or until progression. Treatment with carboplatin+etoposide will continue for a maximum of 4 cycles (up to 2.8 months). Participants who must discontinue 1 of the 2 drugs due to adverse events in the combination may continue the study with the other combination drug.
  Interventions: Drug: Carboplatin; Drug: Etoposide
- Belzutifan (Experimental): Participants with AC mCRPC in Cohort J will receive belzutifan 120mg QD in the initial cohort. If an efficacy signal is detected in this arm based on a totality of evidence, Cohort J may be expanded further where participants will be randomized 1:1 to receive either belzutifan 120 mg QD or belzutifan 120 mg QD and pembrolizumab 200 mg Q3W. Treatment will continue for a maximum of 35 cycles (up to 2 years) or until progression.
  Interventions: Biological: Belzutifan 120mg
- Pembrolizumab+Belzutifan (Experimental): Participants with AC mCRPC in Cohort J will receive belzutifan 120mg QD in the initial cohort. If an efficacy signal is detected in this arm based on a totality of evidence, Cohort J may be expanded further where participants will be randomized 1:1 to receive either belzutifan 120 mg QD or belzutifan 120 mg QD and pembrolizumab 200 mg Q3W. Treatment will continue for a maximum of 35 cycles (up to 2 years) or until progression.
  Interventions: Biological: Pembrolizumab 200 mg; Biological: Belzutifan 120mg

INTERVENTIONS:
Biological: Pembrolizumab 200 mg — IV Q3W
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab+Abiraterone+Prednisone; Pembrolizumab+Belzutifan; Pembrolizumab+Carboplatin+Etoposide; Pembrolizumab+Docetaxel+Prednisone; Pembrolizumab+Enzalutamide; Pembrolizumab+Lenvatinib: AC; Pembrolizumab+Lenvatinib:t-NE; Pembrolizumab+Olaparib
Drug: Olaparib 400 mg — Eight 50-mg capsules PO BID
  Other Names: LYNPARZA®; MK-7339
  Arms: Pembrolizumab+Olaparib
Drug: Docetaxel 75 mg/m^2 — IV Q3W
  Other Names: TAXOTERE®
  Arms: Pembrolizumab+Docetaxel+Prednisone
Drug: Prednisone 5 mg — One 5-mg tablet PO BID
  Arms: Pembrolizumab+Abiraterone+Prednisone; Pembrolizumab+Docetaxel+Prednisone
Drug: Enzalutamide 160 mg — Four 40-mg capsules, four 40-mg tablets, or two 80-mg tablets PO QD
  Other Names: XTANDI®
  Arms: Pembrolizumab+Enzalutamide
Other: Dexamethasone 8 mg — Premedication for Cohort B given PO at 12, 3, and 1 hours prior to docetaxel infusion Q3W
  Arms: Pembrolizumab+Docetaxel+Prednisone
Drug: Olaparib 300 mg — Two 150-mg tablets PO BID
  Other Names: LYNPARZA®; MK-7339
  Arms: Pembrolizumab+Olaparib
Drug: Abiraterone acetate 1000 mg — Two 500-mg or four 250-mg tablets PO QD
  Other Names: ZYTIGA®
  Arms: Pembrolizumab+Abiraterone+Prednisone
Drug: Lenvatinib — 20 mg PO QD
  Other Names: LENVIMA®; MK-7902
  Arms: Pembrolizumab+Lenvatinib: AC; Pembrolizumab+Lenvatinib:t-NE
Biological: Pembrolizumab/Vibostolimab coformulation — IV Q3W
  Other Names: MK-7684A
  Arms: Pembrolizumab/Vibostolimab coformulation; Pembrolizumab/Vibostolimab coformulation:t-NE
Drug: Carboplatin — IV Q3W
  Other Names: PARAPLATIN®
  Arms: Carboplatin+Etoposide; Pembrolizumab+Carboplatin+Etoposide
Drug: Etoposide — IV on Days 1, 2 and 3 of each cycle
  Other Names: TOPOSAR™
  Arms: Carboplatin+Etoposide; Pembrolizumab+Carboplatin+Etoposide
Biological: Belzutifan 120mg — PO QD
  Other Names: WELIREG™
  Arms: Belzutifan; Pembrolizumab+Belzutifan

SUMMARY:
The purpose of this study is to assess the safety and efficacy of pembrolizumab (MK-3475) combination therapy in participants with metastatic castration resistant prostate cancer (mCRPC). There will be ten cohorts in this study: Cohort A will receive pembrolizumab + olaparib, Cohort B will receive pembrolizumab + docetaxel + prednisone, Cohort C will receive pembrolizumab + enzalutamide, Cohort D will receive pembrolizumab + abiraterone + prednisone Cohort E will receive pembrolizumab+lenvatinib, Cohort F will receive pembrolizumab+lenvatinib, Cohort G will receive pembrolizumab/vibostolimab coformulation (MK-7684A), Cohort H will receive pembrolizumab/vibostolimab coformulation, Cohort I will receive pembrolizumab+carboplatin+etoposide in Arm 1 and carboplatin+etoposide in Arm 2 and Cohort J will receive belzutifan in Arm1 and Pembrolizumab+belzutifan in Arm 2. Outcome measures will be assessed individually for each cohort.

DETAILED DESCRIPTION:
Assignment of patients to a cohort will be based on prior treatment as outlined in the eligibility criteria.

Participants who discontinue pembrolizumab or vibostolimab+pembrolizumab after 35 infusions for reasons other than disease progression or intolerability, or who discontinue pembrolizumab or coformulation of pembrolizumab/vibostolimab after attaining a complete response (and had at least 8 administrations of pembrolizumab or pembrolizumab/vibostolimab coformulation and at least 2 treatments with pembrolizumab or pembrolizumab/vibostolimab coformulation beyond initial complete response) may be eligible to receive a second course of treatment that includes up to 17 additional infusions (approximately 1 year) of pembrolizumab monotherapy or pembrolizumab/vibostolimab coformulation after they have experienced radiographic disease progression after stopping first course treatment.

Effective with Protocol Amendment 08, enrollment into Cohorts A, B, C, and D was closed.

Effective with Protocol Amendment 14, enrollment into Cohorts E, F, G, and H was closed (not due to any safety issues). No further efficacy and survival follow-up assessments will be collected in Cohorts A through H.

Effective with Protocol Amendment 16, enrollment into Cohort J was closed (not due to any safety issues).

ELIGIBILITY:
Inclusion Criteria:

* For Cohorts A, B, C, D, E, G, J: Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology

  * For Cohorts F, H, I: Has t-NE or de novo metastatic prostate cancer defined by ≥1% neuroendocrine cells that are located in discrete regions of a recent biopsy specimen from a metastasis as determined by the investigational site and confirmed by central histology review prior to enrollment. Epstein criteria of neuroendocrine differentiation in prostate cancer is used for eligibility. Specimens must have one of the morphologies of Small cell carcinoma or Large cell neuroendocrine carcinoma (LCNEC) or Mixed (small or large cell) NE carcinoma - acinar adenocarcinoma with positive IHC confirmed by central pathology review
* Is able to provide tumor tissue from a site not previously irradiated as follows: Cohorts A, E, G and J: must provide a core or excisional biopsy from soft tissue or bone biopsy within 1 year of screening and after developing mCRPC; Cohort B: must provide an archival tumor tissue sample or tumor tissue from a newly obtained core or excisional biopsy from soft tissue if the lesion is clinically accessible; Cohorts C and D with soft tissue disease: must provide a core or excisional biopsy from a soft tissue lesion if clinically accessible within 1 year of screening and after developing mCRPC and an archival specimen if available; and Cohorts F, H, and I must provide a core or excisional biopsy from soft tissue or a bone biopsy. For de novo metastatic neuroendocrine prostate participants, biopsies must be performed within 1 year of screening. Participants with bone metastasis only must provide an archival tumor tissue specimen
* Has prostate cancer progression within 6 months prior to screening, as determined by the investigator, by means of one of the following: PSA progression as defined by a minimum of 2 rising PSA levels with an interval of ≥1 week between each assessment where the PSA value at screening should be ≥2 ng/mL; radiographic disease progression in soft tissue based on Response Evaluation Criteria In Solid Tumors Version 1.1 criteria with or without PSA progression; radiographic disease progression in bone defined as the appearance of 2 or more new bone lesions on bone scan with or without PSA progression. Participants with de novo neuroendocrine prostate cancer will not need to provide evidence of progression within 6 months
* Has ongoing androgen deprivation with serum testosterone <50 ng/dL (<2.0 nM). Treatment with luteinizing hormone-releasing hormone agonists or antagonists for all cohorts must have been initiated ≥4 weeks prior to first dose of study therapy and must be continued throughout the study. Participants with de novo metastatic NE prostate cancer will not be required to have been previously treated with androgen deprivation therapy (ADT). ADT must be started in these participants by the time of treatment allocation/randomization
* Participants receiving bone resorptive therapy (including, but not limited to bisphosphonate or receptor activator of nuclear factor kappa-β ligand inhibitor) must be on stable doses for ≥4 weeks prior to first dose of study therapy
* Must be abstinent from heterosexual intercourse, refrain from donating sperm, or agree to use contraception (unless confirmed to be azoospermic) during the intervention period starting with the first dose of study therapy. The length of time required to continue contraception after the last dose of study intervention for each study intervention is as follows: 7 days for abiraterone acetate and lenvatinib; 30 days for enzalutamide; and 95 days for olaparib, docetaxel, and carboplatin/etoposide. No contraception measures are required during and after the intervention period for pembrolizumab/vibostolimab coformulation
* Has a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale for Cohorts A and C and a performance status of 0 or 1 for Cohorts B, D, E, F, G, H, I and J within 10 days of study start
* For Cohort A: Has received docetaxel for mCRPC. Prior treatment with 1 other chemotherapy for mCRPC is allowed. Up to 2 second-generation hormonal manipulations (e.g., abiraterone acetate and/or enzalutamide) are allowed. Prior docetaxel for metastatic hormone-sensitive prostate cancer is allowed if ≥4 weeks have elapsed from the last dose of docetaxel prior to day 1 of Cycle 1
* For Cohort B: Has received prior treatment with either abiraterone acetate or enzalutamide (but not both) in the prechemotherapy mCRPC state. Participants in Cohort B must have received at least 4 weeks of either abiraterone or enzalutamide treatment (but not both) who failed treatment or became intolerant of the drug
* For Cohort C: Has received prior treatment with abiraterone acetate in the pre-chemotherapy mCRPC state without prior enzalutamide. Participants in Cohort C must have received at least 4 weeks of abiraterone treatment who failed treatment or become intolerant of the drug. Participants who received abiraterone acetate in the hormone-sensitive state will not be eligible
* For Cohort D: Has not received chemotherapy for mCRPC and has either not had prior second generation hormonal manipulation for mCRPC OR has previously been treated with enzalutamide for mCRPC and failed treatment or has become intolerant of the drug. Prior docetaxel for metastatic hormone-sensitive prostate cancer is allowed if ≥4 weeks have elapsed from the last dose of docetaxel. Prior treatment with abiraterone acetate in the hormone-sensitive metastatic setting is allowed as long as there was no progression on this agent and abiraterone acetate was not discontinued due to adverse events (AEs)
* For Cohorts E, G and J: Has received docetaxel for mCRPC. Prior treatment with 1 other chemotherapy for mCRPC is allowed. Up to 2 second-generation hormonal manipulations (eg, abiraterone acetate, enzalutamide, apalutamide, darolutamide or other next-generation hormonal agents [NHA]) are allowed. Participants who received prior ketoconazole for metastatic disease may be enrolled. If docetaxel chemotherapy is used more than once (eg, once for metastatic hormone-sensitive and once for mCRPC), it will be considered as 1 therapy. Prior docetaxel for metastatic hormone-sensitive prostate cancer (mHSPC) is allowed if ≥4 weeks have elapsed from the last dose of docetaxel prior to Day 1 of Cycle 1
* For Cohort F, H, and I: Participants must have received prior treatment with androgen deprivation therapy (ADT) for metastatic disease. Prior treatment with up to a total of 2 chemotherapies for mCRPC is allowed, as well as up to 2 second-generation hormonal manipulations for mCRPC. Participants who received prior ketoconazole for metastatic disease may be enrolled. Docetaxel for mHSPC is allowed in addition to docetaxel for mCRPC. If docetaxel chemotherapy is used more than once (eg, once for metastatic hormone-sensitive and once for mCRPC), it will be considered as 1 therapy

Exclusion Criteria:

* Has had a prior anticancer monoclonal antibody (mAb) within 4 weeks prior to first dose study therapy or who has not recovered (i.e., Grade ≤1 or at baseline) from AEs due to mAbs administered >4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy abiraterone treatment, enzalutamide treatment, or radiation therapy within 2 weeks prior to first dose of study therapy or who has not recovered (ie, Grade ≤1 or at baseline) from AEs due to a previously administered agent
* Is currently participating in and receiving study therapy or has participated in a study of an investigational agent and received study drug or used an investigational device within 4 weeks of treatment allocation/randomization
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to treatment allocation/randomization
* Has had prior treatment with therapeutic radiopharmaceuticals for prostate cancer, such as Radium-223 or Leutitium-177, within 4 weeks prior to the first dose of trial treatment
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease
* Has previously participated in any other pembrolizumab trial, or received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), and anti-programmed cell death ligand 1 (anti-PD-L2)
* Has a known history of Human Immunodeficiency Virus (HIV)
* Has known active Hepatitis B or Hepatitis C
* Has received a live vaccine or live-attenuated vaccine within 30 days of the first dose of study therapy
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Has a "superscan" bone scan defined as an intense symmetric activity in the bones and diminished renal parenchymal activity on baseline bone scan such that the presence of additional metastases in the future could not be evaluated
* Has had prior solid, organ or bone marrow transplant
* For Cohort A: Has experienced a seizure or seizures within 6 months of study start or is currently being treated with cytochrome P450 enzyme (CYP) inducing anti-epileptic drugs for seizures
* For Cohort A: Is currently receiving strong or moderate inhibitors of CYP3A4 including azole antifungals; macrolide antibiotics; or protease inhibitors
* For Cohort A: Is currently receiving strong or moderate inducers of CYP3A4
* For Cohort A: Has myelodysplastic syndrome
* For Cohort A: Has symptomatic congestive heart failure (New York Heart Association Class III or IV heart disease), unstable angina pectoris, cardiac arrhythmia, or uncontrolled hypertension
* For Cohort B: Has received prior treatment with docetaxel or another chemotherapy agent for metastatic prostate cancer
* For Cohort B: Has peripheral neuropathy Common Terminology Criteria for Adverse Events ≥2 except due to trauma
* For Cohort B: Has ascites and/or clinically significant pleural effusion
* For Cohort B:Has symptomatic congestive heart failure (New York Heart Association Class III or IV heart disease)
* For Cohort B: Is currently receiving any of the following classes of inhibitors of CYP3A4: azole antifungals; macrolide antibiotics; or protease inhibitors
* For Cohort C: Has received prior chemotherapy for mCRPC. Prior docetaxel for metastatic hormone-sensitive prostate cancer is allowed if ≥4 weeks elapsed from last dose of docetaxel. Participants who received abiraterone acetate in the hormone-sensitive state will not be eligible
* For Cohort C: Has a history of seizure or any condition that may predispose to seizure (including, but not limited to prior cerebrovascular accident, transient ischemic attack, or brain arteriovenous malformation; or intracranial masses such as a schwannoma or meningioma that is causing edema or mass effect)
* For Cohort C:Has known or suspected brain metastasis or leptomeningeal carcinomatosis
* For Cohort C: Has a history of loss of consciousness within 12 months of the screening visit
* For Cohort C: Has hypotension (systolic blood pressure <86 millimeters of mercury [mmHg]) or uncontrolled hypertension (systolic blood pressure >170 mmHg or diastolic blood pressure >105 mmHg) at the screening visit
* For Cohort C: Has received treatment with 5-α reductase inhibitors (e.g., finasteride, dutasteride), estrogens, and/or cyproterone within 4 weeks prior to Cycle 1
* For Cohort C: Has a history of prostate cancer progression on ketoconazole
* For Cohort D: Has received prior treatment with docetaxel or another chemotherapy agent for metastatic prostate cancer
* For Cohort D: Has progressed on prior abiraterone acetate for treatment of castration sensitive or resistant metastatic prostate cancer
* For Cohort D: Has discontinued prior treatment with abiraterone acetate due to AEs
* For Cohort D: Has previously been treated with ketoconazole for prostate cancer for >7 days
* For Cohort D: Has received prior systemic treatment with an azole drug (eg, fluconazole, itraconazole) within 4 weeks of Cycle 1, Day 1
* For Cohort D: Has uncontrolled hypertension (systolic BP ≥ 160 mm Hg or diastolic BP ≥ 95 mm Hg)
* For Cohort D: Has a history of pituitary or adrenal dysfunction
* For Cohort D: Has clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association Class II-IV heart disease or cardiac ejection fraction measurement of <50% at baseline
* For Cohort D: Has atrial fibrillation, or other cardiac arrhythmia requiring therapy
* For Cohort D: Has a history of chronic liver disease
* For Cohort D: Is currently receiving strong CYP3A4 inducers (eg, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital) during abiraterone acetate treatment, CYP2D6 substrates with a narrow therapeutic index (for example thioridazine), or CYP2C8 substrates with a narrow therapeutic index (for example pioglitazone)
* For Cohorts E and F: Has a left ventricular ejection fraction (LVEF) below the institutional (or local laboratory) normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO)
* For Cohorts E and F: Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation
* For Cohorts E and F: Has prolongation of QT interval by Fredericia (QTcF) interval to >480 milliseconds
* For Cohorts E and F: Has had major surgery within 3 weeks prior to first dose of study interventions
* For Cohorts E and F: Has pre-existing ≥Grade 3 gastrointestinal or non-gastrointestinal fistula
* For Cohorts E and F: Has had significant cardiovascular impairment within 12 months of the first dose of study intervention, such as history of New York Heart Association >Class II congestive heart failure, unstable angina, myocardial infarction, or cerebrovascular accident (CVA)/stroke, cardiac revascularization procedure, or cardiac arrhythmia associated with hemodynamic instability
* For Cohorts E and F: Has active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of lenvatinib
* For Cohorts E and F: Has gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib
* For Cohorts G, H, and I: Has had a severe hypersensitivity reaction to treatment with another monoclonal antibody
* For Cohorts G, H, and I: Has symptomatic ascites or pleural effusion
* For Cohort I: Has clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, and/or abdominal carcinomatosis
* For Cohort I: Has received previous treatment for prostate cancer with platinum-containing compounds

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be male and be ≥18 years of age on day of signing informed consent.
Enrollment: 1200 (Estimated)
Dates: Start 2016-11-17 (Actual); Primary Completion 2027-10-22 (Estimated); Study Completion 2027-10-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With a Decrease of ≥50% in Prostatic Specific Antigen (PSA) | From Baseline Measured Every 3 Weeks Until Radiographic Progression Estimated to be Approximately 2 Years
Number of Participants with Adverse Events (AEs) | Assessed Every 3 Weeks Over the Duration of the Study Which is Estimated to be Approximately 2 Years
Number of Participants Discontinuing Study Drug Due to AEs | Assessed Every 3 Weeks Over the Duration of the Study Which is Estimated to be Approximately 2 Years
Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed by Blinded Independent Central Review (BICR) | Assessed Over the Duration of the Study Which is Estimated to be Approximately 2 Years

SECONDARY OUTCOMES:
Disease Control Rate (DCR) Based on Prostate Cancer Working Group 3 (PCWG3)-modified RECIST 1.1 Assessed by BICR | Assessed Over the Duration of the Study Which is Estimated to be Approximately 2 Years
Overall Survival (OS) | Assessed Over the Duration of the Study Which is Estimated to be Approximately 2 Years
Duration of Response (DOR) Based on PCWG3-modified RECIST 1.1 Assessed by BICR | Assessed Over the Duration of the Study Which is Estimated to be Approximately 2 Years
ORR Based on PCWG3-modified RECIST 1.1 Assessed by BICR | Assessed Over the Duration of the Study Which is Estimated to be Approximately 2 Years
Time to PSA Progression | Assessed Over the Duration of the Study Which is Estimated to be Approximately 2 Years
Radiographic Progression-free Survival (rPFS) Based on PCWG3-modified RECIST 1.1 Assessed by BICR | Assessed Over the Duration of the Study Which is Estimated to be Approximately 2 Years
Composite Response Rate Defined as Any One of the Following: A. Response Based on RECIST 1.1; B. PSA Decrease of ≥50%; or C. Circulating Tumor-cell Count Conversion (Pembrolizumab + Olaparib Cohort Only) | Assessed Over the Duration of the Study Which is Estimated to be Approximately 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (21):
- United States (7):
  - Call for Information (Investigational Site 2041), Aurora, Colorado
  - Call for Information (Investigational Site 2091), Cleveland, Ohio
  - Call for Information (Investigational Site 2094), Portland, Oregon
  - Call for Information (Investigational Site 0008), Pittsburgh, Pennsylvania
  - Call for Information (Investigational Site 0019), Myrtle Beach, South Carolina
  - Call for Information (Investigational Site 2090), Germantown, Tennessee
  - Call for Information (Investigational Site 0016), Seattle, Washington
- MSD Australia, North Ryde, Australia
- Merck Canada, Kirkland, Quebec, Canada
- MSD Denmark, Glostrup Municipality, Denmark
- MSD France, Paris, France
- MSD Ireland (Human Health) Ltd., Dublin, Ireland
- MSD Italia S.r.l., Rome, Italy
- MSD Comercializadora, S. de R.L. de C.V., Mexico City, Mexico
- Merck Sharp & Dohme BV, Haarlem, Netherlands
- Merck Sharp & Dohme (New Zealand) Ltd.,, Auckland, New Zealand
- MSD Polska Sp. Z o.o., Warsaw, Poland
- Merck Sharp and Dohme de Espana S.A., Madrid, Spain
- MSD Sweden, Stockholm, Sweden
- Merck Sharp & Dohme Ilaclari Ltd. Sti, Istanbul, Turkey (Türkiye)
- Merck Sharp & Dohme Ltd., London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Yu EY, Ferrario C, Linch MD, Stoeckle M, Laguerre B, Arranz JA, Todenhofer T, Fong PC, Piulats JM, Berry W, Emmenegger U, Mourey L, Joshua AM, Mar N, Appleman LJ, Conter HJ, Gravis G, Li XT, Schloss C, Poehlein C, de Bono JS. Pembrolizumab plus Abiraterone Acetate and Prednisone in Patients with Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer: Results from KEYNOTE-365 Cohort D. Eur Urol Oncol. 2025 Jun;8(3):641-651. doi: 10.1016/j.euo.2024.05.013. Epub 2024 Jun 25. PMID 38926066
- [Result] Yu EY, Berry WR, Gurney H, Retz M, Conter HJ, Laguerre B, Fong PCC, Ferrario C, Todenhofer T, Gravis G, Piulats JM, Emmenegger U, Shore ND, Romano E, Mourey L, Li XT, Poehlein CH, Schloss C, Appleman LJ, de Bono JS. Pembrolizumab and Enzalutamide in Patients with Abiraterone Acetate-Pretreated Metastatic Castration-Resistant Prostate Cancer: Cohort C of the Phase 1b/2 KEYNOTE-365 Study. Eur Urol Oncol. 2024 Jun;7(3):509-518. doi: 10.1016/j.euo.2023.10.008. Epub 2023 Nov 7. PMID 37940446
- [Derived] Fong PC, Kwiatkowski M, Mosca A, Valderrama BP, Li C, Huang YH, Zedan AH, Kuc K, Wiechno P, Laguerre B, Gonzalez-Billalabeitia E, Osipov M, Sener Dede D, Goh JC, Daugaard G, Zhu P, Imai K, Liu Y, Arranz Arija JA. Vibostolimab Coformulated with Pembrolizumab in Participants with Docetaxel-pretreated Metastatic Castration-resistant Prostate Cancer: KEYNOTE-365 Cohort G. Eur Urol Focus. 2025 Aug 11:S2405-4569(25)00242-1. doi: 10.1016/j.euf.2025.07.018. Online ahead of print. PMID 40796417
- [Derived] Yu EY, Kolinsky MP, Berry WR, Retz M, Mourey L, Piulats JM, Appleman LJ, Romano E, Gravis G, Gurney H, Bogemann M, Emmenegger U, Joshua AM, Linch M, Sridhar S, Conter HJ, Laguerre B, Massard C, Li XT, Schloss C, Poehlein CH, de Bono JS. Pembrolizumab Plus Docetaxel and Prednisone in Patients with Metastatic Castration-resistant Prostate Cancer: Long-term Results from the Phase 1b/2 KEYNOTE-365 Cohort B Study. Eur Urol. 2022 Jul;82(1):22-30. doi: 10.1016/j.eururo.2022.02.023. Epub 2022 Apr 6. PMID 35397952
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26340&tenant=MT_MSD_9011